CLINICAL TRIAL: NCT07130162
Title: Detection of Phosphatidylinositol Glycan Anchor Biosynthesis Class U Protein as Serum Biomarker for Breast Cancer
Brief Title: Phosphatidylinositol Glycan Anchor Biosynthesis Class U Protein in Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Gamal Neyaz Mohamed, Resident doctor, Assiut University
Other Study IDs: PIGU in breast cancer
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- breast cancer patients: 48 case
  Interventions: Diagnostic Test: Measurement of serum PIGU protein concentrations of patients and controls by Enzyme-Linked Immunosorbent Assay (ELISA)
- healthy controls: 48 case
  Interventions: Diagnostic Test: Measurement of serum PIGU protein concentrations of patients and controls by Enzyme-Linked Immunosorbent Assay (ELISA)

INTERVENTIONS:
Diagnostic Test: Measurement of serum PIGU protein concentrations of patients and controls by Enzyme-Linked Immunosorbent Assay (ELISA) — Measurement of serum PIGU protein concentrations of patients and controls by Enzyme-Linked Immunosorbent Assay (ELISA)

SUMMARY:
The present study aims to evaluate the serum level of PIGU protein in patients with breast cancer and its relation with clinical, laboratory and pathological data of the patients.

DETAILED DESCRIPTION:
Breast cancer (BC) is the most common cancer among females. It is known to be the second leading cause of cancer-related deaths among women worldwide . Although the incidence rates of breast cancer vary between developed and developing nations, it continues to be the most prevalent form of cancer among women in Egypt, with an estimated mortality rate of approximately 11% in 2020 . Breast cancer is a heterogeneous disease, so treatment and prognosis vary based on tumor pathological type, histological grade, lymph node involvement, hormone receptor status and disease stage

* however even patients with similar prognostic features can experience different clinical outcomes after treatment . Despite significant advancements in early screening and diagnostic techniques, the incidence of breast cancer continues to rise annually, accounting for approximately 11.7% of all newly diagnosed cancer cases. So detection of new prognostic indicators is critical for selecting the optimal treatment modalities, evaluating the response and creating a follow-up plan to improve clinical outcome . Phosphatidylinositol glycan anchor biosynthesis class U (PIGU), also known as cell division cycle 91-like 1 (CDC91L1), is an important subunit of glycosylphosphatidylinositol transaminase (GPI-T) complex. It has been reported that the over-activity of certain components of the GPI T complex contributes to the development of various cancers, such as

breast cancer, bladder cancer, lymphoma, and non-small cell lung cancer. Studies have shown that PIGU has the potential to be a prognostic biomarker and therapeutic target for liver cancer, ovarian cancer and colorectal cancer . Also, PIGU expression levels have been associated with radiotherapy for differentiated thyroid cancer and the risk of cutaneous melanoma. It has been demonstrated that PIGU promotes hepatocellular carcinoma (HCC) progression via increasing HCC cell viability, migration, invasion and inhibiting apoptosis by activating the transcription factor nuclear factor-kappa B (NF-κB) pathway . Recent researches verify that PIGU protein levels were significantly higher in breast cancer patients compared to normal people

. So it was speculated that PIGU is playing an important role in tumor development, progression and it can be considered as a marker for breast cancer screening and prognosis (12).

ELIGIBILITY:
Inclusion Criteria:

* The study will be carried on female patients who diagnosed as breast cancer based on pathological and radiological confirmation, recruited from Clinical Oncology Departments and outpatient clinics, SECI, Assiut University

Exclusion Criteria:

* Patients diagnosed with other concomitant cancer.
* Patients who have already received chemotherapy or radiotherapy.

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: female patients who diagnosed as breast cancer based on pathological and radiological confirmation
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Detection of the serum level of PIGU protein in patients with breast cancer | baseline
  Evaluate the relation between serum level of PIGU protein in breast cancer patients and other clinical, laboratory and pathological data of the patients.

REFERENCES:
- [Background] An S, Liu F, Shi Y. Identification of serum phosphatidylinositol glycan anchor biosynthesis class U protein as diagnostic biomarker for breast cancer. Clin Chim Acta. 2025 Mar 1;569:120183. doi: 10.1016/j.cca.2025.120183. Epub 2025 Feb 6. PMID 39922250
- [Background] Giaquinto AN, Sung H, Newman LA, Freedman RA, Smith RA, Star J, Jemal A, Siegel RL. Breast cancer statistics 2024. CA Cancer J Clin. 2024 Nov-Dec;74(6):477-495. doi: 10.3322/caac.21863. Epub 2024 Oct 1. PMID 39352042
- [Background] Azim HA, Elghazawy H, Ghazy RM, Abdelaziz AH, Abdelsalam M, Elzorkany A, Kassem L. Clinicopathologic Features of Breast Cancer in Egypt-Contemporary Profile and Future Needs: A Systematic Review and Meta-Analysis. JCO Glob Oncol. 2023 Mar;9:e2200387. doi: 10.1200/GO.22.00387. PMID 36888929
- [Background] Thakur N, Singh R, Sunigdha, Devgan R, Sharma A. Clinicopathological prognostic factors for survival in patients with breast cancer: a retrospective study from a tertiary cancer centre from North-West India. Ecancermedicalscience. 2025 Mar 6;19:1865. doi: 10.3332/ecancer.2025.1865. eCollection 2025. PMID 40492224
- [Background] Wei X, Yang W, Zhang F, Cheng F, Rao J, Lu L. PIGU promotes hepatocellular carcinoma progression through activating NF-kappaB pathway and increasing immune escape. Life Sci. 2020 Nov 1;260:118476. doi: 10.1016/j.lfs.2020.118476. Epub 2020 Sep 21. PMID 32971102